CLINICAL TRIAL: NCT05765357
Title: Phase I Clinical Study of Randomized, Double-blind, Single-dose, Parallel Comparison of Trastuzumab for Injection and Herceptin® in Healthy Male Volunteers on Pharmacokinetics and Safety
Brief Title: Clinical Study to Compare the Pharmacokinetics and Safety of Trastuzumab for Injection With Herceptin® in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZDTQ-2017-QTZDK
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2017-04

CONDITIONS: Metastatic Breast Cancer; Metastatic Gastric Cancer
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms | interventions — Trastuzumab; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trastuzumab for injection (Experimental): 4mg/kg, Single dose for intravenous infusion
  Interventions: Drug: Trastuzumab for injection
- Herceptin (Active Comparator): 4mg/kg, Single dose for intravenous infusion
  Interventions: Drug: Herceptin

INTERVENTIONS:
Drug: Trastuzumab for injection — Trastuzumab for injection manufactured by Chia Tai Tianqing. Trastuzumab is a humanized IGG1-class monoclonal antibody produced by CHO cells. Its mechanism of action is to prevent the attachment of human epidermal growth factor to Her2 by attaching itself to Her2, thus blocking the growth of cancer cells. In addition, Trastuzumab can also stimulate the body's own immune cells to destroy cancer cells.
  Arms: Trastuzumab for injection
Drug: Herceptin — Herceptin is the brand name of Trastuzumab for injection manufactured by Roche. Trastuzumab is a humanized IGG1-class monoclonal antibody produced by CHO cells. Its mechanism of action is to prevent the attachment of human epidermal growth factor to Her2 by attaching itself to Her2, thus blocking the growth of cancer cells. In addition, Trastuzumab can also stimulate the body's own immune cells to destroy cancer cells.
  Arms: Herceptin

SUMMARY:
Trastuzumab for injection is a biosimilar of Herceptin ® produced by Chia Tai Tianqing Biotechnology Co., LTD, which is a humanized IgG1 monoclonal antibody produced by chinese hamster ovary (CHO) cells. A randomized, double-blind, single-dose, parallel phase I study comparing trastuzumab for injection with Herceptin ® in healthy male volunteers was conducted to evaluate the similarities in pharmacokinetics, tolerability, safety and immunogenicity of Trastuzumab for injection and Herceptin®.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the purpose of the trial, and have a basic understanding of the pharmacological effects and possible adverse reactions of the drug under study; Voluntary written informed consent in accordance with the Helsinki Declaration;
* Healthy male subjects aged ≥ 18 years and ≤ 65 years;
* Body weight ≥ 50 kg ≤ 90 kg, body mass index ≥ 18 ≤ 28kg/m2;
* The system examination indicators were within the normal range, or the examination results were abnormal but the researchers judged that there was no clinical significance;
* Subjects agree to use reliable contraceptive methods for both themselves and their partners during the study period and for 6 months after the study drug infusion.

Exclusion Criteria:

* History of hypertension or abnormal blood pressure at screening/baseline measurement;
* A history of albuminuria or albuminuria as assessed by the investigator as clinically significant;
* Received any antibody or protein targeting Vascular Endothelial Cell Growth Factor (VEGF) or VEGF receptors in the previous 1 year;
* Study the use of any biological product or live virus vaccine within 3 months prior to drug infusion, or the use of any monoclonal antibody within 12 months;
* Have an inherited tendency to bleed or have coagulation dysfunction, or have a history of thrombosis or bleeding;
* History of digestive tract perforation or digestive tract fistula;
* Unhealed wound ulcers or fractures, or major surgery within 2 months prior to randomization or expected to be performed during the study period or within 2 months after study completion;
* Use of a prescription or over-the-counter drug or nutritional supplement within the 5 half-life of the drug or nutritional supplement or within 2 weeks prior to the study drug use;
* Positive virology test;
* Known allergy to trastuzumab;
* Known history of allergic diseases or allergic constitution;
* Study the history of blood donation 3 months before drug infusion;
* Received any other investigational drug therapy or participated in another interventional clinical trial within 2 months prior to screening
* A history of alcohol or drug abuse in the 12 months prior to screening;
* A history of mental illness;
* Subjects whose spouses plan to become pregnant;
* The study cannot be completed according to protocol requirements during the study period;
* Conditions considered unsuitable for inclusion by other researchers.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 89 (Actual)
Dates: Start 2017-07-16 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Area under drug concentration - time curve (AUC0-t) | Within 30 minutes before administration to 1344 hours after administration
  Area under the curve from time zero to the lowest detectable blood drug concentration

SECONDARY OUTCOMES:
Area under drug concentration - time curve (AUC0-∞) | Within 30 minutes before administration to 1344 hours after administration
  The area under the curve extrapolating from time zero to infinity
Peak concentration (Cmax) | Within 30 minutes before administration to 1344 hours after administration
  Peak maximum plasma drug concentration
Time to reach maximum plasma (Tmax) | Within 30 minutes before administration to 1344 hours after administration
  Time to reach maximum plasma concentration after dosing
Clearance (CL) | Within 30 minutes before administration to 1344 hours after administration
  Percentage of the body that eliminates organ-scavenging drugs
half-life (T1/2) | Within 30 minutes before administration to 1344 hours after administration
  The time it takes for serum drug concentrations to drop by half
Apparent volume of distribution (Vd/F) | Within 30 minutes before administration to 1344 hours after administration
  Apparent volume of distribution after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No